CLINICAL TRIAL: NCT06772727
Title: Comparison of Hemodynamic Effect of Lidocaine-based Versus Opioid-based Induction of Anesthesia in Emergency Laparotomy: a Randomized Controlled Trial.
Brief Title: Lidocaine-based Versus Opioid-based Induction of Anesthesia in Emergency Laparotomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MD-265-2024
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Post-induction Hypotension; Lidocaine; Opioid; Emergency Laparotomy
MeSH Terms: interventions — Lidocaine; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Active Comparator): Patients will receive 1 mg/kg lidocaine intravenously (IV)
  Interventions: Drug: Lidocaine; Drug: Propofol; Drug: Succinyl choline
- Fentanyl group (Active Comparator): Patients will receive 1 mcg/kg fentanyl intravenously (IV)
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Succinyl choline

INTERVENTIONS:
Drug: Lidocaine — After preoxygenation with 100% oxygen for 3 minutes, the study drug (lidocaine) will be administered. Patients will receive 1 mg/kg lidocaine of 10 mg/mL lidocaine solution (prepared by diluting 5 mL of lidocaine 20% in saline to a total volume of 10 mL)
  Arms: Lidocaine group
Drug: Fentanyl — After preoxygenation with 100% oxygen for 3 minutes, the study drug (fentanyl) will be administered. Patients will receive 1 mcg/kg fentanyl of 10 mcg/mL fentanyl solution (prepared by diluting 100 mcg fentanyl in saline to a total volume of 10 mL).
  Arms: Fentanyl group
Drug: Propofol — After administration of the study drug, all patients will receive 2 mg/kg propofol intravenously
Drug: Succinyl choline — After loss of consciousness, 1 mg/kg succinyl choline will be administered over 5 seconds, and tracheal intubation will be done through direct laryngoscopy after 60 seconds.

SUMMARY:
The primary role of anesthesia is to provide unconsciousness, amnesia, immobility, and pain control. Other important roles include maintaining stable vital signs and tissue perfusion, preventing and management of organ failure.

Emergency laparotomy represents a major surgical procedure which is usually performed in patients with acute and chronic comorbidities and is associated with several surgical and medical complications with post-induction hypotension being one of the common and serious complication. Thus, it is essential to provide a balanced and safe protocol for anesthesia which maintains adequate hypnosis and antinociception besides vital stability and adequate perfusion.

Opioid drugs are commonly used within the context of balanced general anesthesia primarily for their antinociceptive effects. Opioid drugs had been a basic component of perioperative care for providing analgesia and decreasing the requirements of other hypnotic drugs. However, there are several short- and long-term adverse effects for opioid drugs such as pruritus, postoperative nausea and vomiting, respiratory depression, dependence, and development of chronic pain. Furthermore, opioid drugs are claimed to have cardiovascular depressant effects which increases the risk of hypotension if they were used routinely in patients with borderline hemodynamic profile. Therefore, there is an increased interest in opioid-sparing and opioid-free anesthesia and several international consensus statements were released to regulate and suggest protocols for opioid-sparing anesthetic regimens.

Lidocaine-based anesthesia had been recently reported as a successful regimen for induction of anesthesia in elderly population with better hemodynamic profile than opioid-based induction. The investigators hypothesize that lidocaine-based induction of anesthesia would provide superior hemodynamic profile compared to conventional opioid-based induction of anesthesia in emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Both gender
3. American Society of Anesthesiologists (ASA) class I-III undergoing emergency laparotomy.

Exclusion Criteria:

1. Patient refusal
2. Severe cardiac morbidities (impaired contractility with ejection fraction < 45%, heart block, arrhythmias, tight valvular lesions)
3. Baseline mean arterial pressure <75 mmHg
4. Patients on vasopressor infusion,
5. Patients with high shock index (heart rate / systolic blood pressure >1)
6. Pregnant or lactating women,
7. Allergy of any of the study drugs
8. Hypertensive patients and patients on beta blockers.
9. Uncontrolled hypertensive patients or patients receiving angiotensin converting enzyme (ACE) inhibitors preoperatively.
10. Opioid drug abusers.
11. Patients with increased intracranial tension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension | immediately after induction of anesthesia until 20 minutes after induction of anesthesia
  Incidence of post-induction hypotension

SECONDARY OUTCOMES:
Norepinephrine dose | from induction of anesthesia until 20 minutes after skin incision
  Total norepinephrine dose during the period from induction of anesthesia until 20-minutes after intubation or skin incision
Heart rate | every 2 minutes for 20 minutes after induction of anesthesia
Mean Arterial Pressure | every 2 minutes for 20 minutes after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jehan Elkholy, M.D., Study Chair — Cairo University; Eman F Ali,, M.D., Study Director — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University; Mohsen M Waheeb, M.D., Study Director — Cairo University; Samar M Abdel Azeim Ghazala, M.Sc., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt